CLINICAL TRIAL: NCT01719627
Title: PILOT STUDY OF PROTECTION AGAINST ex Vivo HIV INFECTION IN RECTAL MUCOSA IN HEALTHY VOLUNTEERS AFTER ADMINISTRATION OF MARAVIROC
Brief Title: First Study to Evaluate the Capacity of Maraviroc Drug to Protect Against HIV Infection in Samples of Rectal Mucosa From Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Fundación FLS de Lucha Contra el Sida, las Enfermedades Infecciosas y la Promoción de la Salud y la Ciencia (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: MARAVIPREX
Record Dates: First submitted 2012-10-10; First posted 2012-11-01 (Estimated); Last update posted 2015-03-05 (Estimated); Status verified 2015-03

CONDITIONS: HIV
Keywords: HIV, Maraviroc, PrEP, Ex vivo infection, rectal mucosa.
MeSH Terms: interventions — Maraviroc

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- MVC 300 mg (Experimental): MVC 300 mg in unique dose
  Interventions: Drug: Maraviroc
- TVD 300/200 QD (Active Comparator): TVD 300/200 QD during 7 days.
  Interventions: Drug: TVD 300/200 QD
- Maraviroc 600mg (Experimental): MVC 600mg in unique dose
  Interventions: Drug: Maraviroc

INTERVENTIONS:
Drug: Maraviroc — Unique dose of Maraviroc 300mg
  Arms: MVC 300 mg
Drug: TVD 300/200 QD — TVD 300/200 QD during 7 days
  Arms: TVD 300/200 QD
Drug: Maraviroc — Unique dose of Maraviroc 600mg
  Arms: Maraviroc 600mg

SUMMARY:
Pre-exposure prophylaxis (PrEP) is a method of preventing HIV infection through the use of antiretroviral (ARV) medications before exposure to HIV. This study will assess the potential of MVC as a "on demand" pre-exposure prophylaxis, within a strategy for the prevention of HIV infection in men who have sex with men (MSM).

DETAILED DESCRIPTION:
Several clinical trials are currently under way evaluating the safety and effectiveness of ARV-based PrEP for preventing HIV infection. The results of the first efficacy trials of ARV-based PrEP showed fewer HIV infections among study participants receiving the study drugs compared to those receiving placebo. Although the results are promising, concerns about adherence, pharmacokinetics, and toxicity still needs further exploration so new and more effective preventive pharmacological approaches should be evaluated. This trial will evaluate the safety, pharmacokinetics and efficacy of ex vivo HIV infection of rectal mucosa by the CCR5 antagonist drug maraviroc (Selzentry) administered to healthy volunteers. This trial will last approximately one year. Twenty-one volunteers will receive MVC 300 mg orally in a single dose. Study visits will occur at enrollment and at days 0, 7, 9, 14 and 16. All study visits will include a physical examination, blood collection and storage and in the basal visit and a day 7 or 9 the participants will undergo a colonoscopy. Ex vivo HIV infectivity in rectal mucosa biopsies and plasma/mucosa MVC levels will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

1. Men who have sex with men (MSM)
2. Age 18 years or above
3. HIV negative at the time of inclusion 4. Signed informed consent

Exclusion Criteria:

1. Existence of sexually transmitted infection (STI) or active systemic infection
2. Submit a contraindication to rectal biopsy
3. Take any drugs concomitantly with interactions with the MVC
4. Subject unable to follow protocol

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2012-10; Primary Completion 2014-05 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Infectivity of HIV: p24 production | Baseline
  HIV replication will be measured by the determination of HIV p24 production in culture supernatant after 12 days of culture. The HIV production in ex vivo cultures from the basal and after drug administration will be compared and the results will be expressed as a measure of Maraviroc efficacy.
Infectivity of HIV: p24 production | Visit 1 (Group 1: day 8, Group 2: day 7, Grop 3: day 9)
  HIV replication will be measured by the determination of HIV p24 production in culture supernatant after 12 days of culture. The HIV production in ex vivo cultures from the basal and after drug administration will be compared and the results will be expressed as a measure of Maraviroc efficacy.

SECONDARY OUTCOMES:
Maraviroc plasmatic levels | Visit 1 (Group 1: day 8, Group 2: day 7, Grop 3: day 9)
Maraviroc levels in rectal mucosa | Visit 1 (Group 1: day 8, Group 2: day 7, Grop 3: day 9)
Truvada plasmatic levels | Visit 1 (day 7)
Truvada levels in rectal mucosa | Visit 1 (day 7)

CONTACTS AND LOCATIONS:
Locations (1):
- Germans Trias i Pujol Hospital, Badalona, Barcelona, Spain